CLINICAL TRIAL: NCT03637764
Title: A Phase 1/2 Open-label, Multi-center, Safety, Preliminary Efficacy and Pharmacokinetic (PK) Study of Isatuximab (SAR650984) in Combination With Atezolizumab or Isatuximab Alone in Patients With Advanced Malignancies
Brief Title: Safety, Preliminary Efficacy and PK of Isatuximab (SAR650984) Alone or in Combination With Atezolizumab in Patients With Advanced Malignancies
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was stopped after interim analysis for 4 cohorts (HCC, SCCHN, EOC, and GBM) indicated that the results did not fulfill the preplanned interim analysis criteria to move to Phase 2 stage 2 in all 4 cohorts.
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACT15377; 2018-000390-67 (EudraCT Number); U1111-1202-0839 (Other: UTN)
Record Dates: First submitted 2018-08-05; First posted 2018-08-20 (Actual); Results first posted 2023-06-08 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-05

CONDITIONS: Neoplasm
Keywords: Anti-CD38 monoclonal antibody
MeSH Terms: conditions — Neoplasms | interventions — isatuximab; atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort A: HCC: Isatuximab + Atezolizumab (Experimental): Participants with hepatocellular carcinoma (HCC) received atezolizumab 1200 milligrams, every 3 weeks (Q3W), intravenous (IV) infusion along with isatuximab 10 milligrams per kilogram (mg/kg), IV infusion, once weekly for 3 weeks (i.e., on Day 1, Day 8 and Day 15 of Cycle 1) and then Q3W (i.e., on Day 1 of each 21- day treatment cycle) until disease progression, unacceptable adverse events (AE), participant's decision to stop the treatment, or death or study cut-off whichever occurred first (maximum duration of exposure: 106 weeks).
  Interventions: Drug: Isatuximab SAR650984; Drug: Atezolizumab
- Cohort B: SCCHN: Isatuximab + Atezolizumab (Experimental): Participants with squamous cell carcinoma of the head and neck (SCCHN) received atezolizumab 1200 milligrams,Q3W, IV infusion along with isatuximab 10 mg/kg, IV infusion, once weekly for 3 weeks (i.e., on Day 1, Day 8 and Day 15 of Cycle 1) and then Q3W (i.e., on Day 1 of each 21- day treatment cycle) until disease progression, unacceptable AE, participant's decision to stop the treatment, or death or study cut-off whichever occurred first (maximum duration of exposure: 108 weeks).
  Interventions: Drug: Isatuximab SAR650984; Drug: Atezolizumab
- Cohort C: EOC: Isatuximab + Atezolizumab (Experimental): Participants with epithelial ovarian cancer (EOC) received atezolizumab 1200 mg, Q3W, IV infusion along with isatuximab 10 mg/kg, IV infusion, once weekly for 3 weeks (i.e., on Day 1, Day 8 and Day 15 of Cycle 1) and then Q3W (i.e., on Day 1 of each 21- day treatment cycle) until disease progression, unacceptable AE, participant's decision to stop the treatment, or death or study cut-off whichever occurred first (maximum duration of exposure: 61 weeks).
  Interventions: Drug: Isatuximab SAR650984; Drug: Atezolizumab
- Cohort D-1: GBM: Isatuximab + Atezolizumab (Experimental): Participants with glioblastoma multiforme (GBM) received atezolizumab 1200 mg, Q3W, IV infusion along with isatuximab 10 mg/kg, IV infusion, once weekly for 3 weeks (i.e., on Day 1, Day 8 and Day 15 of Cycle 1) and then Q3W (i.e., on Day 1 of each 21- day treatment cycle) until disease progression, unacceptable AE, participant's decision to stop the treatment, or death or study cut-off whichever occurred first (maximum duration of exposure: 54 weeks).
  Interventions: Drug: Isatuximab SAR650984; Drug: Atezolizumab

INTERVENTIONS:
Drug: Isatuximab SAR650984 — Pharmaceutical form: solution for infusion
  Route of administration: intravenous
  Other Names: Sarclisa
Drug: Atezolizumab — Pharmaceutical form: solution for infusion
  Route of administration: intravenous
  Other Names: Tecentriq®

SUMMARY:
Primary Objectives:

* Phase 1: To characterize the safety and tolerability of isatuximab in combination with atezolizumab in participants with unresectable hepatocellular carcinoma (HCC), platinum-refractory recurrent/metastatic squamous cell carcinoma of the head and neck (SCCHN), platinum-resistant/refractory epithelial ovarian cancer (EOC), or recurrent glioblastoma multiforme (GBM), and to determine the recommended Phase 2 dose (RP2D).
* Phase 2: To assess response rate (RR) of isatuximab in combination with atezolizumab in participants with HCC or SCCHN or EOC.
* Phase 2: To assess the progression free survival rate at 6 months (PFS-6) of isatuximab in combination with atezolizumab, or as a single agent in participants with GBM.

Secondary Objectives:

* To evaluate the safety profile of isatuximab monotherapy (GBM only), or in combination with atezolizumab in Phase 2.
* To evaluate the immunogenicity of isatuximab and atezolizumab.
* To characterize the pharmacokinetic (PK) profile of isatuximab single agent (GBM only) and atezolizumab in combination with isatuximab.
* To assess the overall efficacy of isatuximab in combination with atezolizumab, or single agent (GBM only).

DETAILED DESCRIPTION:
The total study duration per participant was up to 28 months including up to 28 days screening period, up to 24 months treatment period, and a 3 month safety follow up period.

ELIGIBILITY:
Inclusion criteria:

* Participants must have a known diagnosis of either unresectable HCC, platinum-refractory recurrent/metastatic SCCHN, platinum-resistant/refractory EOC with evidence of measurable disease or recurrent GBM.
* Greater than or equal to (>=)18 years of age.
* For participants with HCC: Documentation of progressive disease (PD) during or after treatment with either sorafenib or lenvatinib, or intolerance to the therapy.
* For participants with SCCHN: Received and failed up to 2 lines of prior systemic anti-cancer therapy with documentation of tumor recurrence or PD within 6 months of last platinum-based therapy in primary, recurrent, or metastatic setting.
* For participants with EOC: Received up to 3 lines of prior platinum-containing therapy when the disease was platinum-sensitive, and the participants should not have received any systemic therapy for platinum-resistant/refractory disease. Specific to France only: Documentation of PD on or after 1 line of anti-cancer therapy for platinum resistant/refractory disease (unless participants are ineligible or intolerant to standard of care for platinum-resistant/refractory disease).
* For participants with GBM: Documentation of PD or first recurrence during or after temozolomide maintenance therapy for newly diagnosed GBM treated with 1st line radiotherapy plus concurrent temozolomide.

Exclusion criteria:

* Prior exposure to agent that blocks CD38 or participation in clinical studies with isatuximab.
* For participants with HCC, SCCHN, EOC or GBM prior exposure to any agent (approved or investigational) that blocks the PD-1/PD-L1 pathway.
* Evidence of other immune related disease /conditions.
* History of non-infectious pneumonitis requiring steroids or current pneumonitis; history of the thoracic radiation.
* Received a live-virus vaccination within 28 days of planned treatment start. Seasonal flu vaccines that do not contain live virus are permitted.
* Prior solid organ or bone marrow transplantation.
* Eastern Cooperative Oncology Group performance status >=2 for participants with HCC, SCCHN or EOC or Karnofsky performance score less than or equal to (<=) 70 for participants with GBM.
* Poor bone marrow reserve.
* Poor organ function.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2022-05-11 (Actual); Study Completion 2022-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (26):
- United States (3):
  - Investigational Site Number :8400004, Santa Monica, California
  - Investigational Site Number :8400007, Boston, Massachusetts
  - Investigational Site Number :8400002, Houston, Texas
- Belgium (2):
  - Investigational Site Number :0560001, Brussels
  - Investigational Site Number :0560002, Ghent
- Investigational Site Number :1240001, Toronto, Ontario, Canada
- Czechia (3):
  - Investigational Site Number :2030001, Brno
  - Investigational Site Number :2030003, Olomouc
  - Investigational Site Number :2030002, Prague
- Italy (4):
  - Investigational Site Number :3800007, Meldola, Forlì-Cesena
  - Investigational Site Number :3800003, Rozzano, Milano
  - Investigational Site Number :3800009, Milan
  - Investigational Site Number :3800004, Padua
- Investigational Site Number :5280001, Rotterdam, Netherlands
- Spain (6):
  - Investigational Site Number :7240001, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number :7240006, Hospitalet de Llobregat, Castille and León
  - Investigational Site Number :7240004, Madrid, Madrid, Comunidad de
  - Investigational Site Number :7240003, Madrid / Madrid, Madrid, Comunidad de
  - Investigational Site Number :7240008, Pamplona, Navarre
  - Investigational Site Number :7240007, Madrid
- Taiwan (6):
  - Investigational Site Number :1580005, Kaohsiung City
  - Investigational Site Number :1580002, Tainan
  - Investigational Site Number :1580003, Taipei
  - Investigational Site Number :1580006, Taipei
  - Investigational Site Number :1580004, Taipei
  - Investigational Site Number :1580001, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Background] Simonelli M, Garralda E, Eskens F, Gil-Martin M, Yen CJ, Obermannova R, Chao Y, Lonardi S, Melichar B, Moreno V, Yu ML, Bongiovanni A, Calvo E, Rottey S, Machiels JP, Gonzalez-Martin A, Paz-Ares L, Chang CL, Mason W, Lin CC, Reardon DA, Vieito M, Santoro A, Meng R, Abbadessa G, Menas F, Lee H, Liu Q, Combeau C, Ternes N, Ziti-Ljajic S, Massard C. Isatuximab plus atezolizumab in patients with advanced solid tumors: results from a phase I/II, open-label, multicenter study. ESMO Open. 2022 Oct;7(5):100562. doi: 10.1016/j.esmoop.2022.100562. Epub 2022 Aug 18. PMID 35987165

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 26 active sites in 8 countries. A total of 107 participants were enrolled between 06 August 2018 and 21 July 2020 and received isatuximab in combination with atezolizumab. Study was planned to be conducted in 2 parts: Phase 1 (safety run-in) and Phase 2 (efficacy with a 2-stage design).
Pre-assignment Details: Study was stopped after performance of interim analysis for 4 cohorts (Cohort A [HCC], Cohort B [SCCHN], Cohort C [EOC] & Cohort D-1 [GBM]) indicated that efficacy results observed in each cohort did not fulfill the preplanned interim analysis criteria allowing the study to move to Phase 2 Stage 2 in these 4 cohorts. Participant flow, Baseline, outcome measures and safety data were analyzed on combined Phase 1 and 2 populations.
Groups:
- Cohort A: Hepatocellular Carcinoma (HCC): Isatuximab + Atezolizumab: Participants with hepatocellular carcinoma (HCC) received atezolizumab 1200 milligrams (mg), every 3 weeks (Q3W), intravenous (IV) infusion along with isatuximab 10 milligrams per kilogram (mg/kg), IV infusion, once weekly for 3 weeks (i.e., on Day 1, Day 8 and Day 15 of Cycle 1) and then Q3W (i.e., on Day 1 of each 21- day treatment cycle) until disease progression, unacceptable adverse events (AE), participant's decision to stop the treatment, or death or study cut-off whichever occurred first (maximum duration of exposure: 106 weeks).
- Cohort B: Squamous Cell Carcinoma of the Head and Neck (SCCHN): Isatuximab + Atezolizumab: Participants with squamous cell carcinoma of the head and neck (SCCHN) received atezolizumab 1200 milligrams,Q3W, IV infusion along with isatuximab 10 mg/kg, IV infusion, once weekly for 3 weeks (i.e., on Day 1, Day 8 and Day 15 of Cycle 1) and then Q3W (i.e., on Day 1 of each 21- day treatment cycle) until disease progression, unacceptable AE, participant's decision to stop the treatment, or death or study cut-off whichever occurred first (maximum duration of exposure: 108 weeks).
- Cohort C: Epithelial Ovarian Cancer (EOC): Isatuximab + Atezolizumab: Participants with epithelial ovarian cancer (EOC) received atezolizumab 1200 mg, Q3W, IV infusion along with isatuximab 10 mg/kg, IV infusion, once weekly for 3 weeks (i.e., on Day 1, Day 8 and Day 15 of Cycle 1) and then Q3W (i.e., on Day 1 of each 21- day treatment cycle) until disease progression, unacceptable AE, participant's decision to stop the treatment, or death or study cut-off whichever occurred first (maximum duration of exposure: 61 weeks).
- Cohort D-1: Glioblastoma Multiforme (GBM): Isatuximab + Atezolizumab: Participants with glioblastoma multiforme (GBM) received atezolizumab 1200 mg, Q3W, IV infusion along with isatuximab 10 mg/kg, IV infusion, once weekly for 3 weeks (i.e., on Day 1, Day 8 and Day 15 of Cycle 1) and then Q3W (i.e., on Day 1 of each 21- day treatment cycle) until disease progression, unacceptable AE, participant's decision to stop the treatment, or death or study cut-off whichever occurred first (maximum duration of exposure: 54 weeks).
Period: Overall Study
Arm/Group | Cohort A: Hepatocellular Carcinoma (HCC): Isatuximab + Atezolizumab | Cohort B: Squamous Cell Carcinoma of the Head and Neck (SCCHN): Isatuximab + Atezolizumab | Cohort C: Epithelial Ovarian Cancer (EOC): Isatuximab + Atezolizumab | Cohort D-1: Glioblastoma Multiforme (GBM): Isatuximab + Atezolizumab
Started | 27 | 29 | 18 | 33
Completed (Participants who completed the study treatment duration.) | 1 | 3 | 0 | 0
Not Completed | 26 | 26 | 18 | 33
Not completed — Adverse Event | 2 | 0 | 0 | 1
Not completed — Progressive Disease | 23 | 23 | 18 | 31
Not completed — Withdrawal by Subject | 1 | 3 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all-treated population that included all the participants who signed the study informed consent and received at least 1 dose of the study treatments, either isatuximab or atezolizumab.
Groups:
- Cohort A: HCC: Isatuximab + Atezolizumab: Participants with HCC received atezolizumab 1200 mg, Q3W, IV infusion along with isatuximab 10 mg/kg, IV infusion, once weekly for 3 weeks (i.e., on Day 1, Day 8 and Day 15 of Cycle 1) and then Q3W (i.e., on Day 1 of each 21- day treatment cycle) until disease progression, unacceptable AE, participant's decision to stop the treatment, or death or study cut-off whichever occurred first (maximum duration of exposure: 106 weeks).
- Cohort B: SCCHN: Isatuximab + Atezolizumab: Participants with SCCHN received atezolizumab 1200 mg, Q3W, IV infusion along with isatuximab 10 mg/kg, IV infusion, once weekly for 3 weeks (i.e., on Day 1, Day 8 and Day 15 of Cycle 1) and then Q3W (i.e., on Day 1 of each 21- day treatment cycle) until disease progression, unacceptable AE, participant's decision to stop the treatment, or death or study cut-off whichever occurred first (maximum duration of exposure: 108 weeks).
- Cohort C: EOC: Isatuximab + Atezolizumab: Participants with EOC received atezolizumab 1200 mg, Q3W, IV infusion along with isatuximab 10 mg/kg, IV infusion, once weekly for 3 weeks (i.e., on Day 1, Day 8 and Day 15 of Cycle 1) and then Q3W (i.e., on Day 1 of each 21- day treatment cycle) until disease progression, unacceptable AE, participant's decision to stop the treatment, or death or study cut-off whichever occurred first (maximum duration of exposure: 61 weeks).
- Cohort D-1: GBM: Isatuximab + Atezolizumab: Participants with GBM received atezolizumab 1200 mg, Q3W, IV infusion along with isatuximab 10 mg/kg, IV infusion, once weekly for 3 weeks (i.e., on Day 1, Day 8 and Day 15 of Cycle 1) and then Q3W (i.e., on Day 1 of each 21- day treatment cycle) until disease progression, unacceptable AE, participant's decision to stop the treatment, or death or study cut-off whichever occurred first (maximum duration of exposure:54 weeks).
- Total: Total of all reporting groups
Arm/Group | Cohort A: HCC: Isatuximab + Atezolizumab | Cohort B: SCCHN: Isatuximab + Atezolizumab | Cohort C: EOC: Isatuximab + Atezolizumab | Cohort D-1: GBM: Isatuximab + Atezolizumab | Total
Number analyzed (Participants) | 27 | 29 | 18 | 33 | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (11.8) | 61.1 (9.1) | 56.3 (10.6) | 53.3 (13.3) | 58.3 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 18 | 10 | 38
  Male | 20 | 26 | 0 | 23 | 69
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 11 | 9 | 4 | 0 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 15 | 20 | 13 | 29 | 77
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLTs: AEs occurring during 1st treatment cycle, unless due to disease progression/obviously unrelated cause which included: hematological abnormalities: Grade(G) 4 neutropenia(N) for 7 or more consecutive days, G3 to G4 N with fever (temperature greater than or equal to [>=] 38.5 degree Celsius on more than 1 occasion) or microbiologically/radiographically documented infection, G3 thrombocytopenia with clinically significant bleeding/ G4 thrombocytopenia. Non-hematological abnormalities: G >=2 Aspartate transaminase (AST)/ Alanine transaminase (ALT) elevation simultaneous with G >=2 total bilirubin elevation without initial findings of cholestasis or any other reason found, G4 non-hematologic AE, G3 to 4 cytokine release syndrome, G3 non-hematological AE lasting greater than (>)3 days, delay in initiation of Cycle 2 >14 days due to treatment related laboratory abnormalities/AE. Any other AE that study committee deemed to be dose-limiting, regardless of grade, was also considered DLT.
Time Frame: Cycle 1 (21 days)
Population: Analysis was performed on DLT evaluable population that included participants who received planned doses of isatuximab and atezolizumab during Cycle 1 and who completed the DLT observation period.
Measure: Count of Participants; unit: Participants
Groups:
- Isatuximab + Atezolizumab: Participants with HCC, SCCHN, EOC, or GBM received atezolizumab 1200 mg, Q3W, IV infusion along with isatuximab 10 mg/kg, IV infusion, once weekly for 3 weeks (i.e., on Day 1, Day 8 and Day 15 of Cycle 1) and then Q3W (i.e., on Day 1 of each 21- day treatment cycle) until disease progression, unacceptable AE, participant's decision to stop the treatment, or death or study cut-off whichever occurred first.
Arm/Group | Isatuximab + Atezolizumab
Number analyzed (Participants) | 9
Participants | 0

2. Primary Outcome: Recommended Phase 2 Dose (RP2D)
Description: RP2D was the starting dose selected for Phase 2 part of the study. RP2D was the selected dose at which no more than 1 out of 6 participants (starting dose or dose level minus -1 [DL-1]) or 2 out of 12 participants (starting dose) experienced a DLT related to the investigational medicinal product. DLTs: Adverse Event (AE) occurring during 1st treatment cycle, unless due to disease progression/obviously unrelated cause included: hematological abnormalities: G4 N for 7/ more consecutive days, G3 to G4 N with fever, G3/G4 thrombocytopenia. Non-hematological abnormalities: G>=2 AST/ALT elevation simultaneous with G >=2 total bilirubin elevation without cholestasis or any other reason found, G4 non-hematologic AE, G3 to 4 cytokine release syndrome, G3 non-hematological AE lasting >3 days, delay in initiation of Cycle 2 >14 days due to treatment related laboratory abnormalities/AE.
Time Frame: Cycle 1 (21 days)
Population: Analysis was performed on DLT evaluable population.
Measure: Number; unit: milligrams per kilogram (mg/kg)
Arm/Group | Isatuximab + Atezolizumab
Number analyzed (Participants) | 9
milligrams per kilogram (mg/kg) | 10

3. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: MTD was defined as the highest dose level at which no more than 1 out of 6 participants (starting dose or DL-1) or 2 out of 12 participants (starting dose) experienced a DLT related to the investigational medicinal product. DLTs: AE occurring during 1st treatment cycle, unless due to disease progression/obviously unrelated cause included: hematological abnormalities: G4 N for 7 or more consecutive days, G3 to G4 N with fever, G3 or G4 thrombocytopenia. Non-hematological abnormalities: G>=2 AST/ ALT elevation simultaneous with G >=2 total bilirubin elevation without cholestasis or any other reason found, G4 non-hematologic AE, G3 to 4 cytokine release syndrome, G3 non-hematological AE lasting >3 days, delay in initiation of Cycle 2 >14 days due to treatment related laboratory abnormalities or AEs.
Time Frame: Cycle 1 (21 days)
Population: Analysis was performed on DLT evaluable population.
Measure: Number; unit: mg/kg
Arm/Group | Isatuximab + Atezolizumab
Number analyzed (Participants) | 9
mg/kg | 10

4. Primary Outcome: Percentage of Participants With Overall Response (OR): For HCC/SCCHN/EOC Cohorts
Description: OR was defined as the percentage of participants with complete response (CR) and partial response (PR) as best overall response, assessed per RECIST 1.1 criteria. Best overall response was derived per RECIST 1.1 criteria using disease assessments performed from the first dose of treatment throughout the study excluding any assessments performed after the cut-off date or following the initiation of a further anticancer treatment. CR was defined as the disappearance of all target lesions, pathological lymph nodes (target/non-target)- reduction in short axis <10 mm; PR was defined as at least 30% decrease in sum of diameters of target lesions, taking as reference baseline sum diameters. Disease progression was defined as at least a 20% increase in sum of diameters of target lesions, taking as reference smallest sum, sum with an absolute increase of diameter of at least 5 mm and appearance of >1 new lesion.
Time Frame: From randomization until disease progression, or death or study cut-off whichever occurred first (maximum duration of exposure: up to 108 weeks)
Population: Analysis was performed on all-treated population. Data for this outcome measure was not planned to be collected and analyzed for GBM Cohort as pre-specified in protocol.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: HCC: Isatuximab + Atezolizumab | Cohort B: SCCHN: Isatuximab + Atezolizumab | Cohort C: EOC: Isatuximab + Atezolizumab
Number analyzed (Participants) | 27 | 29 | 18
percentage of participants | 7.4 [1.3 to 21.5] | 13.8 [4.9 to 28.8] | 5.6 [0.3 to 23.8]

5. Primary Outcome: Probability of Participants With Progression Free Survival at 6 Months (PFS-6): GBM Cohort
Description: PFS-6 was defined as the probability of participants alive without disease progression at 6 months as assessed by RANO criteria. Participants who didn't experience documented progression or death before analysis cut-off date or date of initiation of new anticancer treatment, PFS was censored at date of last valid disease assessment not showing progression performed prior to initiation of further anticancer treatment or analysis cut-off date, whichever was 1st. Per RANO criteria, progressive disease was defined as >=25% increase size of T1- gadolinium enhancing disease, or increased T2/FLAIR signal, or presence of new lesion, or worsening clinical status. PFS-6 was evaluated by Kaplan-Meier method.
Time Frame: From randomization until 6 months after the last participant's first treatment in the GBM Cohort D-1
Population: Analysis was performed on all-treated population. Data for this outcome measure was not planned to be collected and analyzed for Cohorts A: HCC, Cohort B: SCCHN and Cohort C: EOC as pre-specified in protocol.
Measure: Number (95% Confidence Interval); unit: probability of participants
Groups:
- Cohort D-1: GBM: Isatuximab + Atezolizumab: Participants with GBM received atezolizumab 1200 mg, Q3W, IV infusion along with isatuximab 10 mg/kg, IV infusion, once weekly for 3 weeks (i.e., on Day 1, Day 8 and Day 15 of Cycle 1) and then Q3W (i.e., on Day 1 of each 21- day treatment cycle) until disease progression, unacceptable AE, participant's decision to stop the treatment, or death or study cut-off whichever occurred first (maximum duration of exposure: 54 weeks).
Arm/Group | Cohort D-1: GBM: Isatuximab + Atezolizumab
Number analyzed (Participants) | 33
probability of participants | 0.033 [0.002 to 0.145]

6. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Treatment-emergent Adverse Events (TESAEs)
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug and did not necessarily have to have a causal relationship with the treatment. Serious adverse events (SAEs) were any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a medically important event. TEAEs were defined as AEs that developed, worsened or became serious during the TEAE period (defined as the time from the first dose of study treatment up to 30 days after the last dose of study treatment).
Time Frame: From Baseline up to 30 days after last study treatment administration (maximum duration of exposure: 106 weeks for Cohort A, 108 weeks for Cohort B, 61 weeks for Cohort C and 54 weeks for Cohort D-1)
Population: Analysis was performed on all-treated population.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: HCC: Isatuximab + Atezolizumab | Cohort B: SCCHN: Isatuximab + Atezolizumab | Cohort C: EOC: Isatuximab + Atezolizumab | Cohort D-1: GBM: Isatuximab + Atezolizumab
Number analyzed (Participants) | 27 | 29 | 18 | 33
Participants
  TEAE | 26 | 29 | 18 | 33
  TESAE | 12 | 16 | 8 | 9

7. Primary Outcome: Number of Participants With Hematological Abnormalities
Description: Hematological parameters assessed were anemia, white blood cell (WBC) decreased, platelet count decreased, lymphocyte count decreased, and neutrophil count decreased. Parameters were assessed as per the National Cancer Institute Common Terminology Criteria for Adverse Experience version 4.03, where Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Potentially Life Threatening. Grade refers to the severity of the AEs.
Time Frame: as for outcome 6
Population: Analysis was performed on all-treated population. Here, 'overall number of participants analyzed' signifies participants with available data for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: HCC: Isatuximab + Atezolizumab | Cohort B: SCCHN: Isatuximab + Atezolizumab | Cohort C: EOC: Isatuximab + Atezolizumab | Cohort D-1: GBM: Isatuximab + Atezolizumab
Number analyzed (Participants) | 26 | 29 | 18 | 32
Participants
  Anemia: Grade 1 | 11 | 13 | 6 | 7
  Anemia: Grade 2 | 5 | 12 | 6 | 2
  Anemia: Grade 3 | 2 | 3 | 0 | 0
  Anemia: Grade 4 | 0 | 0 | 0 | 0
  White blood cell decreased: Grade 1 | 9 | 5 | 4 | 12
  White blood cell decreased: Grade 2 | 2 | 1 | 2 | 3
  White blood cell decreased: Grade 3 | 0 | 0 | 1 | 0
  White blood cell decreased: Grade 4 | 0 | 0 | 0 | 0
  Platelet count decreased: Grade 1 | 11 | 5 | 5 | 10
  Platelet count decreased: Grade 2 | 1 | 0 | 0 | 0
  Platelet count decreased: Grade 3 | 1 | 1 | 0 | 0
  Platelet count decreased: Grade 4 | 1 | 0 | 0 | 0
  Lymphocyte count decreased: Grade 1 | 4 | 2 | 2 | 10
  Lymphocyte count decreased: Grade 2 | 8 | 14 | 7 | 12
  Lymphocyte count decreased: Grade 3 | 3 | 7 | 4 | 3
  Lymphocyte count decreased: Grade 4 | 0 | 4 | 0 | 1
  Neutrophil count decreased: Grade 1 | 3 | 1 | 0 | 1
  Neutrophil count decreased: Grade 2 | 0 | 0 | 3 | 2
  Neutrophil count decreased: Grade 3 | 0 | 0 | 0 | 0
  Neutrophil count decreased: Grade 4 | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Participants With Abnormal Electrolyte Parameters
Description: Electrolyte parameters assessed were hyponatremia, hypernatremia, hypokalemia, hyperkalemia, hypocalcemia, hypercalcemia, hypoalbuminemia, hypoglycemia and hyperglycemia. Parameters were assessed as per the National Cancer Institute Common Terminology Criteria for Adverse Experience version 4.03, where Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Potentially Life Threatening. Grade refers to the severity of the AEs.
Time Frame: as for outcome 6
Population: Analysis was performed on all-treated population. Here 'overall number of participants analyzed' signifies participants with available data for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: HCC: Isatuximab + Atezolizumab | Cohort B: SCCHN: Isatuximab + Atezolizumab | Cohort C: EOC: Isatuximab + Atezolizumab | Cohort D-1: GBM: Isatuximab + Atezolizumab
Number analyzed (Participants) | 26 | 29 | 18 | 32
Participants
  Hyponatremia: Grade 1 | 9 | 12 | 8 | 4
  Hyponatremia: Grade 2 | 0 | 0 | 0 | 0
  Hyponatremia: Grade 3 | 1 | 4 | 0 | 1
  Hyponatremia: Grade 4 | 0 | 0 | 0 | 0
  Hypokalemia: Grade 1 | 2 | 5 | 4 | 4
  Hypokalemia: Grade 2 | 0 | 0 | 0 | 0
  Hypokalemia: Grade 3 | 0 | 2 | 0 | 0
  Hypokalemia: Grade 4 | 0 | 0 | 0 | 0
  Hyperkalemia: Grade 1 | 5 | 6 | 2 | 2
  Hyperkalemia: Grade 2 | 1 | 0 | 1 | 1
  Hyperkalemia: Grade 3 | 0 | 0 | 0 | 0
  Hyperkalemia: Grade 4 | 0 | 0 | 0 | 0
  Hypocalcemia: Grade 1 | 9 | 7 | 2 | 9
  Hypocalcemia: Grade 2 | 0 | 0 | 0 | 0
  Hypocalcemia: Grade 3 | 0 | 0 | 0 | 0
  Hypocalcemia: Grade 4 | 0 | 0 | 0 | 0
  Hypercalcemia: Grade 1 | 1 | 5 | 0 | 0
  Hypercalcemia: Grade 2 | 0 | 2 | 0 | 0
  Hypercalcemia: Grade 3 | 1 | 2 | 0 | 0
  Hypercalcemia: Grade 4 | 0 | 1 | 0 | 0
  Hypoalbuminemia: Grade 1 | 9 | 7 | 7 | 2
  Hypoalbuminemia: Grade 2 | 1 | 3 | 1 | 1
  Hypoalbuminemia: Grade 3 | 0 | 2 | 0 | 0
  Hypoalbuminemia: Grade 4 | 0 | 0 | 0 | 0
  Hypoglycemia: Grade 1 | 1 | 3 | 0 | 2
  Hypoglycemia: Grade 2 | 1 | 0 | 0 | 0
  Hypoglycemia: Grade 3 | 0 | 0 | 0 | 0
  Hypoglycemia: Grade 4 | 0 | 0 | 0 | 0
  Hyperglycemia: Grade 1 | 10 | 7 | 2 | 8
  Hyperglycemia: Grade 2 | 5 | 6 | 2 | 0
  Hyperglycemia: Grade 3 | 1 | 0 | 0 | 2
  Hyperglycemia: Grade 4 | 0 | 1 | 0 | 0
  Hypernatremia: Grade 1 | 0 | 4 | 0 | 5
  Hypernatremia: Grade 2 | 0 | 0 | 0 | 0
  Hypernatremia: Grade 3 | 0 | 0 | 0 | 0
  Hypernatremia: Grade 4 | 0 | 0 | 0 | 0

9. Primary Outcome: Number of Participants With Renal Function Abnormalities
Description: Abnormal renal parameters assessed were creatinine clearance (CrCl), creatinine increased and hyperuricemia. Creatinine clearance was assessed in categories: >=60 - less than (<) 90 milliliters per minute per 1.73 square meter (mL/min/1.73m^2), >=30 - <60 mL/min/1.73m^2, >=15 - <30 mL/min/1.73m^2 and <15 mL/min/1.73m^2. Parameters were assessed as per the National Cancer Institute Common Terminology Criteria for Adverse Experience version 4.03, where Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Potentially Life Threatening. Grade refers to the severity of the AEs.
Time Frame: as for outcome 6
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: HCC: Isatuximab + Atezolizumab | Cohort B: SCCHN: Isatuximab + Atezolizumab | Cohort C: EOC: Isatuximab + Atezolizumab | Cohort D-1: GBM: Isatuximab + Atezolizumab
Number analyzed (Participants) | 26 | 29 | 18 | 32
Participants
  CrCl: >=60 - <90 mL/min/1.73m^2 | 8 | 13 | 10 | 16
  CrCl: >=30 - <60mL/min/1.73m^2 | 5 | 4 | 5 | 1
  CrCl: >=15 - <30 mL/min/1.73m^2 | 3 | 0 | 0 | 0
  CrCl: <15 mL/min/1.73m^2 | 0 | 1 | 0 | 0
  Creatinine increased: Grade 1 | 22 | 19 | 13 | 24
  Creatinine increased: Grade 2 | 2 | 2 | 2 | 0
  Creatinine increased: Grade 3 | 1 | 1 | 0 | 0
  Creatinine increased: Grade 4 | 0 | 0 | 0 | 0
  Hyperuricemia: Grade 1 | 0 | 0 | 0 | 0
  Hyperuricemia: Grade 2 | 0 | 0 | 0 | 0
  Hyperuricemia: Grade 3 | 5 | 7 | 5 | 3
  Hyperuricemia: Grade 4 | 1 | 1 | 1 | 0

10. Primary Outcome: Number of Participants With Liver Abnormalities
Description: Abnormal liver function parameters assessed were AST increased, ALT increased, alkaline phosphatase (ALP) increased, blood bilirubin (BB) increased. Parameters were assessed as per the National Cancer Institute Common Terminology Criteria for Adverse Experience version 4.03, where Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Potentially Life Threatening. Grade refers to the severity of the AEs.
Time Frame: as for outcome 6
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: HCC: Isatuximab + Atezolizumab | Cohort B: SCCHN: Isatuximab + Atezolizumab | Cohort C: EOC: Isatuximab + Atezolizumab | Cohort D-1: GBM: Isatuximab + Atezolizumab
Number analyzed (Participants) | 26 | 29 | 18 | 32
Participants
  AST increased: Grade 1 | 14 | 5 | 6 | 3
  AST increased: Grade 2 | 5 | 0 | 0 | 1
  AST increased: Grade 3 | 3 | 0 | 0 | 0
  AST increased: Grade 4 | 1 | 0 | 0 | 0
  ALT increased: Grade 1 | 11 | 8 | 6 | 11
  ALT increased: Grade 2 | 4 | 0 | 1 | 0
  ALT increased: Grade 3 | 2 | 0 | 0 | 1
  ALT increased: Grade 4 | 1 | 0 | 0 | 0
  ALP increased: Grade 1 | 12 | 13 | 7 | 0
  ALP increased: Grade 2 | 8 | 2 | 3 | 0
  ALP increased: Grade 3 | 2 | 0 | 1 | 0
  ALP increased: Grade 4 | 0 | 0 | 0 | 0
  BB increased: Grade 1 | 6 | 1 | 0 | 0
  BB increased: Grade 2 | 2 | 0 | 0 | 2
  BB increased: Grade 3 | 3 | 0 | 0 | 0
  BB increased: Grade 4 | 1 | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Anti-drug Antibodies (ADA) Response Against Isatuximab
Description: ADA responses were categorized as treatment boosted ADA and treatment-induced ADA. Treatment boosted ADA was defined as pre-existing ADAs with a significant increase in the ADA titer during the study compared to the Baseline titer. Treatment-induced ADA was defined as ADA that developed at any time during the ADA on-study observation period in participants without pre-existing ADA (including participants without pretreatment samples).
Time Frame: From Baseline up to 30 days after last study treatment administration (maximum duration of exposure:106 weeks for Cohort A, 108 weeks for Cohort B, 61 weeks for Cohort C and 54 weeks for Cohort D-1)
Population: Analysis was performed on ADA evaluable population which included all participants who received at least 1 dose of study treatment with at least 1 non-missing ADA result after the drug administration. Here 'overall number of participants analyzed' signifies participants with available data for this outcome measure.
Measure: Number; unit: count of participants
Arm/Group | Cohort A: HCC: Isatuximab + Atezolizumab | Cohort B: SCCHN: Isatuximab + Atezolizumab | Cohort C: EOC: Isatuximab + Atezolizumab | Cohort D-1: GBM: Isatuximab + Atezolizumab
Number analyzed (Participants) | 25 | 24 | 17 | 30
count of participants
  Treatment-induced ADA | 2 | 0 | 1 | 1
  Treatment boosted ADA | 0 | 0 | 0 | 0

12. Secondary Outcome: Number of Participants With Anti-drug Antibodies (ADA) Response Against Atezolizumab
Description: as for outcome 11
Time Frame: as for outcome 6
Population: Analysis was performed on ADA evaluable population. Here 'overall number of participants analyzed' signifies participants with available data for this outcome measure.
Measure: Number; unit: count of participants
Arm/Group | Cohort A: HCC: Isatuximab + Atezolizumab | Cohort B: SCCHN: Isatuximab + Atezolizumab | Cohort C: EOC: Isatuximab + Atezolizumab | Cohort D-1: GBM: Isatuximab + Atezolizumab
Number analyzed (Participants) | 25 | 25 | 17 | 30
count of participants
  Treatment-induced ADA | 2 | 2 | 1 | 0
  Treatment boosted ADA | 0 | 0 | 0 | 0

13. Secondary Outcome: Pharmacokinetics (PK): Maximum Concentration Observed (Cmax) After the First Infusion of Isatuximab
Description: Cmax was defined as the maximum concentration observed after the first administration calculated using the noncompartmental analysis after the intravenous infusion of isatuximab.
Time Frame: At start of infusion (SOI), end of infusion (EOI), EOI+4 hours, 72 hours and 168 hours post-dose on Day 1 of Cycle 1
Population: Analysis was performed on PK population which included all participants who received at least 1 dose of the study treatment with at least one reportable concentration after the study drug administration.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | Cohort A: HCC: Isatuximab + Atezolizumab | Cohort B: SCCHN: Isatuximab + Atezolizumab | Cohort C: EOC: Isatuximab + Atezolizumab | Cohort D-1: GBM: Isatuximab + Atezolizumab
Number analyzed (Participants) | 25 | 26 | 16 | 28
micrograms per milliliter (mcg/mL) | 219 (50.5) | 218 (48.7) | 262 (69.7) | 266 (66.7)

14. Secondary Outcome: Pharmacokinetics (PK): Concentration Observed at the End of Intravenous Infusion (Ceoi) of Isatuximab
Description: Ceoi is the plasma concentration observed at the end of intravenous infusion of isatuximab.
Time Frame: At end of infusion on Cycle 1 Day 1
Population: Analysis was performed on PK population.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Cohort A: HCC: Isatuximab + Atezolizumab | Cohort B: SCCHN: Isatuximab + Atezolizumab | Cohort C: EOC: Isatuximab + Atezolizumab | Cohort D-1: GBM: Isatuximab + Atezolizumab
Number analyzed (Participants) | 25 | 26 | 16 | 28
mcg/mL | 216 (50.8) | 207 (54.9) | 251 (77.3) | 263 (68.8)

15. Secondary Outcome: Pharmacokinetics (PK): Time to Reach Cmax (Tmax) After First Infusion of Isatuximab
Description: Tmax was defined as the time to reach Cmax, calculated using the non-compartmental analysis after the intravenous infusion of isatuximab.
Time Frame: At SOI, EOI, EOI+4 hours, 72 hours and 168 hours post-dose on Day 1 of Cycle 1
Population: Analysis was performed on PK population.
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort A: HCC: Isatuximab + Atezolizumab | Cohort B: SCCHN: Isatuximab + Atezolizumab | Cohort C: EOC: Isatuximab + Atezolizumab | Cohort D-1: GBM: Isatuximab + Atezolizumab
Number analyzed (Participants) | 25 | 26 | 16 | 28
hours | 4.00 [2.42 to 7.92] | 3.37 [2.08 to 8.95] | 6.83 [3.00 to 8.83] | 4.13 [2.65 to 8.38]

16. Secondary Outcome: Pharmacokinetics (PK): Last Concentration Observed Above the Lower Limit of Quantification (Clast) After the First Infusion of Isatuximab
Description: Clast was defined as the last concentration of isatuximab observed above the lower limit of quantification.
Time Frame: At SOI, EOI, EOI+4 hours, 72 hours and 168 hours post-dose on Day 1 of Cycle 1
Population: Analysis was performed on PK population.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Cohort A: HCC: Isatuximab + Atezolizumab | Cohort B: SCCHN: Isatuximab + Atezolizumab | Cohort C: EOC: Isatuximab + Atezolizumab | Cohort D-1: GBM: Isatuximab + Atezolizumab
Number analyzed (Participants) | 25 | 26 | 16 | 28
mcg/mL | 75.9 (35.3) | 67.8 (20.4) | 86.0 (22.2) | 103 (28.4)

17. Secondary Outcome: Pharmacokinetics (PK): Time of Clast (Tlast) After First Infusion of Isatuximab
Description: Tlast was defined as the time of last concentration observed above the lower limit of quantification, calculated using the non-compartmental analysis after the intravenous infusion of isatuximab.
Time Frame: At SOI, EOI, EOI+4 hours, 72 hours and 168 hours post-dose on Day 1 of Cycle 1
Population: Analysis was performed on PK population.
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort A: HCC: Isatuximab + Atezolizumab | Cohort B: SCCHN: Isatuximab + Atezolizumab | Cohort C: EOC: Isatuximab + Atezolizumab | Cohort D-1: GBM: Isatuximab + Atezolizumab
Number analyzed (Participants) | 25 | 26 | 16 | 28
hours | 166 [75.4 to 191] | 167 [162 to 192] | 167 [152 to 212] | 166 [136 to 192]

18. Secondary Outcome: Pharmacokinetics (PK): Area Under the Plasma Concentration Time Curve From Time 0 to Last Quantifiable Concentration (AUClast) After First Infusion of Isatuximab
Description: AUClast was defined as area under the plasma concentration versus time curve calculated from time 0 to last quantifiable concentration. AUClast was calculated using the non-compartmental analysis after the intravenous infusion of isatuximab.
Time Frame: At SOI, EOI, EOI+4 hours, 72 hours and 168 hours post-dose on Day 1 of Cycle 1
Population: Analysis was performed on PK population.
Measure: Mean (Standard Deviation); unit: micrograms*hour/milliliter (mcg*h/mL)
Arm/Group | Cohort A: HCC: Isatuximab + Atezolizumab | Cohort B: SCCHN: Isatuximab + Atezolizumab | Cohort C: EOC: Isatuximab + Atezolizumab | Cohort D-1: GBM: Isatuximab + Atezolizumab
Number analyzed (Participants) | 25 | 26 | 16 | 28
micrograms*hour/milliliter (mcg*h/mL) | 20000 (4570) | 19700 (4500) | 24400 (7120) | 26300 (6510)

19. Secondary Outcome: Pharmacokinetics (PK): Area Under the Plasma Concentration Time Curve Over the Dosing Interval (AUC0-168h) After First Infusion of Isatuximab
Description: AUC0-168h was defined as the area under the plasma concentration versus time curve from time 0 to 168 hours post dose calculated using non-compartmental analysis after first infusion of isatuximab.
Time Frame: At SOI, EOI, EOI+4 hours, 72 hours and 168 hours post-dose on Day 1 of Cycle 1
Population: Analysis was performed on PK population.
Measure: Mean (Standard Deviation); unit: mcg*h/mL
Arm/Group | Cohort A: HCC: Isatuximab + Atezolizumab | Cohort B: SCCHN: Isatuximab + Atezolizumab | Cohort C: EOC: Isatuximab + Atezolizumab | Cohort D-1: GBM: Isatuximab + Atezolizumab
Number analyzed (Participants) | 25 | 26 | 16 | 28
mcg*h/mL | 20200 (4510) | 19800 (4590) | 24300 (6500) | 26400 (6270)

20. Secondary Outcome: Pharmacokinetics (PK): Trough Plasma Concentrations (Ctrough) of Isatuximab
Description: Ctrough was the plasma concentration of isatuximab observed just before treatment administration during repeated dosing.
Time Frame: Pre-infusion on Cycle 1 Day 1, Cycle 1 Day 8 and Cycle 1 Day 15
Population: Analysis was performed on participants who received at least 1 dose of the study treatment with at least one reportable concentration after drug administration; and were ADA negative (i.e., participants without any treatment induced or treatment boosted ADA-positive sample during the treatment or follow-up observation period). Here 'Number analyzed' signifies participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Cohort A: HCC: Isatuximab + Atezolizumab | Cohort B: SCCHN: Isatuximab + Atezolizumab | Cohort C: EOC: Isatuximab + Atezolizumab | Cohort D-1: GBM: Isatuximab + Atezolizumab
Number analyzed (Participants) | 14 | 16 | 10 | 19
mcg/mL
  Cycle 1 Day 1: number analyzed (Participants) | 12 | 10 | 6 | 19
  Cycle 1 Day 1 | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Cycle 1 Day 8: number analyzed (Participants) | 14 | 16 | 10 | 14
  Cycle 1 Day 8 | 67.4 (20.0) | 71.0 (25.9) | 88.6 (21.8) | 99.9 (26.9)
  Cycle 1 Day 15: number analyzed (Participants) | 13 | 15 | 8 | 19
  Cycle 1 Day 15 | 153 (46.8) | 121 (25.6) | 176 (33.6) | 231 (102)

21. Secondary Outcome: Plasma Concentration of Atezolizumab
Time Frame: Cycle 1 Day 1, Cycle 2 Day 1, Cycle 3 Day 1, Cycle 4 Day 1, Cycle 8 Day 1 and Cycle 16 Day 1
Population: Data for the plasma concentration of atezolizumab is not reported because no sample was collected after study termination and analyzed as the study did not fulfil the predefined criteria for Atezolizumab PK analysis.
Groups:
- Cohort A: HCC: Isatuximab + Atezolizumab: Participants with HCC received atezolizumab 1200 mg, Q3W, IV infusion along with isatuximab 10 mg/kg, IV infusion, once weekly for 3 weeks (i.e., on Day 1, Day 8 and Day 15 of Cycle 1) and then Q3W (i.e., on Day 1 of each 21- day treatment cycle) until disease progression, unacceptable AE, participant's decision to stop the treatment, or death or study cut-off whichever occurred first (maximum duration of exposure:106 weeks).
- Cohort B: SCCHN: Isatuximab + Atezolizumab: Participants with SCCHN received atezolizumab 1200 mg, Q3W, IV infusion along with isatuximab 10 mg/kg, IV infusion, once weekly for 3 weeks (i.e., on Day 1, Day 8 and Day 15 of Cycle 1) and then Q3W (i.e., on Day 1 of each 21- day treatment cycle) until disease progression, unacceptable AE, participant's decision to stop the treatment, or death or study cut-off whichever occurred first (maximum duration of exposure:108 weeks).
Arm/Group | Cohort A: HCC: Isatuximab + Atezolizumab | Cohort B: SCCHN: Isatuximab + Atezolizumab | Cohort C: EOC: Isatuximab + Atezolizumab | Cohort D-1: GBM: Isatuximab + Atezolizumab
Number analyzed (Participants) | 0 | 0 | 0 | 0

22. Secondary Outcome: Best Percent Change From Baseline in Tumor Burden
Description: Best tumor burden change was defined as the best percent-change from baseline in a sum of the diameters (longest for non-nodal lesion, short axis for nodal lesions) for all target lesions.
Time Frame: From randomization until progression or death or study cut-off date whichever occurred first (maximum duration of exposure: up to 108 weeks)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Cohort A: HCC: Isatuximab + Atezolizumab | Cohort B: SCCHN: Isatuximab + Atezolizumab | Cohort C: EOC: Isatuximab + Atezolizumab | Cohort D-1: GBM: Isatuximab + Atezolizumab
Number analyzed (Participants) | 25 | 21 | 17 | 24
percent change | 6.2 (31.5) | -3.4 (41.6) | 16.2 (51.1) | 196.6 (347.5)

23. Secondary Outcome: Percentage of Participants With Disease Control (DC) >=6 Months
Description: DC: percentage of participants with complete response (CR), partial response (PR) & stable disease (SD) rate. RANO criteria, CR: no change in size of T1-gadolinium-enhancing (T1-Gd+) disease, stable/ reduced (red) T2/FLAIR signal, no new lesion (NL), no corticosteroid use (CU) & stable/ red clinical status (CS); PR: >=50% change in size of T1-Gd+ disease, stable/red T2/FLAIR signal, no NL, stable/ red CU & stable/ improved CS (ICS). SD: <50% reduction to <25% increase (inc) size of T1-Gd+ disease, stable/red T2/FLAIR signal, no NL, stable/red CU & stable/ICS. Progressive disease (PD): >=25% inc size of T1-Gd+ disease/ inc T2/FLAIR signal/ presence of NL/ worsening CS. RECIST criteria: CR: Disappearance of target lesions. Reduction in short axis to <10 mm of lymph nodes; PR: 30% decrease in sum of diameters of target lesions; PD: 20% inc in sum of diameters of target lesions; SD: Neither sufficient shrinkage from baseline study to qualify for PR nor sufficient inc to qualify for PD.
Time Frame: From the date of first response to disease progression or death, or study cut-off whichever occurred first (maximum duration of exposure: up to 108 weeks)
Population: Analysis was performed on all-treated population.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: HCC: Isatuximab + Atezolizumab | Cohort B: SCCHN: Isatuximab + Atezolizumab | Cohort C: EOC: Isatuximab + Atezolizumab | Cohort D-1: GBM: Isatuximab + Atezolizumab
Number analyzed (Participants) | 27 | 29 | 18 | 33
percentage of participants | 37.0 [21.7 to 54.7] | 41.4 [25.9 to 58.3] | 33.3 [15.6 to 55.4] | 3.0 [0.2 to 13.6]

24. Secondary Outcome: Duration of Response (DOR)
Description: Time from date of 1st response until date of first documented recurrent/progressive disease (PD) or death whichever occurred 1st. In absence of disease progression or death before analysis cut-off date or date of initiation of further anticancer treatment, DOR was censored at date of last valid response. RECIST 1.1 criteria was used for assessment in HCC/SCCHN/EOC Cohorts and RANO criteria for GBM Cohort. Per RECIST 1.1, CR: disappearance of all target lesions; PR: at least 30% decrease in sum of diameters of target lesions, PD: at least 20% increase in sum of diameters of target lesions. Per RANO criteria; CR: no change in size of T1-Gd+ disease, stable/reduced T2/FLAIR signal, no new lesion, no corticosteroid use, and stable/improved status; PR: >=50% change in size of T1-Gd+, stable/reduced T2/FLAIR signal, no new lesion, stable/reduced corticosteroid use, and stable/improved status. PD:>=25% increase size of T1-Gd+/increased T2/FLAIR signal/presence of new lesion/worsening status.
Time Frame: From the date of first response until disease progression or death, or study cut-off date whichever occurred first (maximum duration of exposure: up to 108 weeks)
Population: Analysis was performed on all treated population. Here 'overall number of participants analyzed' signifies participants with available data for this outcome measure and '0' in 'overall number of participants analyzed' signifies that no participant in the Cohort D-1 achieved any response, and hence, no DOR was analyzed.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Cohort A: HCC: Isatuximab + Atezolizumab | Cohort B: SCCHN: Isatuximab + Atezolizumab | Cohort C: EOC: Isatuximab + Atezolizumab | Cohort D-1: GBM: Isatuximab + Atezolizumab
Number analyzed (Participants) | 2 | 4 | 1 | 0
months | 7.5 (3.0) | 20.6 (7.3) | 10.4 |

25. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as time (in months) from 1st study treatment administration to date of 1st documented radiographic progression or date of death from any cause, whichever was 1st. Participants who didn't experience progression or death before analysis cut-off date/date of initiation of new anticancer treatment, PFS was censored at date of last valid disease assessment not showing progression performed prior to initiation of further anticancer treatment or analysis cut-off date, whichever was 1st. RECIST 1.1 criteria was used for assessment in HCC/SCCHN/EOC Cohorts and RANO criteria for GBM Cohort. Per RECIST 1.1 criteria, PD: at least 20% increase in sum of diameters of target lesions, taking as reference smallest sum on study. Appearance of 1 or more new lesions was also considered progression. Per RANO criteria, PD: >=25% increase in product of perpendicular diameters of any target lesion, or worsening neurologic status not explained by causes unrelated to tumor progression.
Time Frame: From date of first study treatment administration until disease progression or death or study cut-off whichever occurred first (maximum duration of exposure: up to 108 weeks)
Population: Analysis was performed on all-treated population. Kaplan-Meier method was used for analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A: HCC: Isatuximab + Atezolizumab | Cohort B: SCCHN: Isatuximab + Atezolizumab | Cohort C: EOC: Isatuximab + Atezolizumab | Cohort D-1: GBM: Isatuximab + Atezolizumab
Number analyzed (Participants) | 27 | 29 | 18 | 33
months | 2.04 [1.840 to 4.008] | 2.10 [1.873 to 3.253] | 2.04 [1.906 to 3.943] | 1.28 [1.216 to 1.380]

26. Secondary Outcome: Percentage of Participants With Response as Per Response Assessment for Neuro-Oncology (RANO) Criteria: GBM Cohort
Description: Response rate for participants with GBM was defined as percentage of participants with CR & PR as best overall response (BOR), assessed by Investigators using RANO criteria. BOR was derived per RANO criteria using disease assessments performed from 1st dose of treatment through study excluding any assessments performed after cut-off date or following initiation of further anticancer treatment. Per RANO criteria; CR was defined as no change in size of T1-gadolinium-enhancing (T1-Gd+) disease, stable or reduced T2/FLAIR signal, no new lesion, no corticosteroid use, and stable or improved clinical status; PR was defined as >=50% change in size of T1-Gd+ disease, stable or reduced T2/FLAIR signal, no new lesion, stable or reduced corticosteroid use, and stable or improved clinical status. Progressive disease was defined as >=25% increase size of T1-Gd+ disease, or increased T2/FLAIR signal, or presence of new lesion, or worsening clinical status.
Time Frame: From randomization until progression, or death, or study cut-off whichever occurred first (maximum duration of exposure: 54 weeks for Cohort D-1)
Population: Analysis was performed on all-treated population. Data for this outcome measure was not collected and analyzed for Cohort A, B and C because the RANO criteria for the assessment of response could not be used to assess the response for solid tumors such as HCC, SCCHN and EOC.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort D-1: GBM: Isatuximab + Atezolizumab
Number analyzed (Participants) | 33
percentage of participants | 0 [0.0 to 8.7]

ADVERSE EVENTS:
Time Frame: From Baseline up to 30 days after last study treatment administration (maximum duration of exposure: 106 weeks for Cohort A, 108 weeks for Cohort B, 61 weeks for Cohort C and 54 weeks for Cohort D-1)
Description: Analysis was performed on all-treated population.
Arm/Group | Cohort A: HCC: Isatuximab + Atezolizumab | Cohort B: SCCHN: Isatuximab + Atezolizumab | Cohort C: EOC: Isatuximab + Atezolizumab | Cohort D-1: GBM: Isatuximab + Atezolizumab
All-Cause Mortality (participants affected / at risk) | 4/27 | 8/29 | 3/18 | 1/33
Serious Adverse Events (participants affected / at risk) | 12/27 | 16/29 | 8/18 | 9/33
Other Adverse Events (participants affected / at risk) | 25/27 | 24/29 | 18/18 | 32/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: HCC: Isatuximab + Atezolizumab (N=27) | Cohort B: SCCHN: Isatuximab + Atezolizumab (N=29) | Cohort C: EOC: Isatuximab + Atezolizumab (N=18) | Cohort D-1: GBM: Isatuximab + Atezolizumab (N=33)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Localised Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periorbital Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia Bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyuria (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant Ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin Neoplasm Bleeding (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour Associated Fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour Rupture (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral Motor Neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Status Epilepticus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arterial Haemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Laryngeal Oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoperitoneum (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intra-Abdominal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Immune-Mediated Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck Mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal Failure (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disease Progression (General disorders) | 3 (3) | 4 (4) | 3 (3) | 1 (1)
General Physical Health Deterioration (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood Bilirubin Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood Creatinine Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Euthanasia (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device Occlusion (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: HCC: Isatuximab + Atezolizumab (N=27) | Cohort B: SCCHN: Isatuximab + Atezolizumab (N=29) | Cohort C: EOC: Isatuximab + Atezolizumab (N=18) | Cohort D-1: GBM: Isatuximab + Atezolizumab (N=33)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Ear Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (5) | 0 (0) | 1 (2) | 0 (0)
Oral Herpes (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (2) | 2 (3) | 2 (2) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Tumour Associated Fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Lymph Node Pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Adrenal Insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 6 (6) | 2 (2) | 3 (3) | 1 (1)
Confusional State (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Disturbance In Attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 4 (4)
Headache (Nervous system disorders) | 3 (3) | 4 (4) | 1 (1) | 12 (18)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Motor Dysfunction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Tremor (Nervous system disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Dry Eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periorbital Oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Visual Acuity Reduced (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear Pruritus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Diastolic Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hot Flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (3)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 4 (4)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 4 (4) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Abdominal Distension (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 6 (10) | 0 (0) | 4 (4) | 2 (2)
Abdominal Pain Lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 3 (3) | 0 (0) | 3 (3) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (5) | 5 (5) | 1 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 3 (4) | 5 (5) | 4 (4)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (7) | 4 (4) | 5 (6) | 3 (3)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (3) | 4 (5) | 4 (5)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Onycholysis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 3 (3) | 1 (1)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 2 (2) | 2 (2)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Asthenia (General disorders) | 3 (3) | 6 (7) | 6 (6) | 8 (8)
Catheter Site Haematoma (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 5 (5) | 6 (6) | 7 (7) | 7 (8)
Non-Cardiac Chest Pain (General disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Oedema Peripheral (General disorders) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
Pyrexia (General disorders) | 3 (5) | 7 (10) | 3 (3) | 1 (1)
Vessel Puncture Site Haemorrhage (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Platelet Count Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Weight Decreased (Investigations) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 16 (17) | 9 (9) | 14 (15) | 17 (18)

LIMITATIONS AND CAVEATS:
Study was stopped after performance of interim analysis for 4 cohorts (Cohort A [HCC], Cohort B [SCCHN], Cohort C [EOC] & Cohort D-1 [GBM]) as the efficacy results observed in each cohort did not fulfill the pre-planned interim analysis criteria allowing the study to move to Phase 2 Stage 2 in these 4 cohorts.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2020-11-23): https://cdn.clinicaltrials.gov/large-docs/64/NCT03637764/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-12): https://cdn.clinicaltrials.gov/large-docs/64/NCT03637764/SAP_001.pdf